CLINICAL TRIAL: NCT06098365
Title: The Effects of Cervical Stabilization Exercises and Isometric Cervical Exercises on Pain, Strength, Flexibility, Disability and Quality of Life in Patients With Cervical Disc Herniation
Brief Title: The Effects of CSE and ISE on Pain, Strength, Flexibility, Disability and QoL in Patients With CDH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, osman coban, Asst. Prof., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UskudaruniversityU
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cervical Disc Herniation
Keywords: Cervical Disc Herniation; stabilization exercises; isometric exercises; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Stabilization Exercise Group (Experimental): After applying traditional treatment for 40 minutes to the cases in Group A, additional segmental cervical stabilization exercises (20 minutes) will be applied.
  Interventions: Other: segmental cervical stabilization exercises
- Cervical Isometric Exercise Group (Other): After applying traditional treatment for 40 minutes to the cases in Group B, additional cervical isometric exercises (20 minutes) will be applied.
  Interventions: Other: cervical isometric exercises

INTERVENTIONS:
Other: segmental cervical stabilization exercises — Segmental spine stabilization exercises were composed of axial extension, cervical extension exercises, cervico-scapulothoracic strengthening and cranio-cervical flexion exercises.
  Other Names: Traditional physiotherapy treatment (40 minutes)
  Arms: Cervical Stabilization Exercise Group
Other: cervical isometric exercises — Cervical isometric exercises consist of 6 sets in a sitting position, each movement lasting 10 seconds, each repeated 5 times, with a 5-second rest in between.
  Other Names: Traditional physiotherapy treatment (40 minutes)
  Arms: Cervical Isometric Exercise Group

SUMMARY:
Cervical disc herniation is a common source of cervical radiculopathy, which can occur suddenly due to trauma and results from chemical and mechanical degenerative changes that occur over time, with an annual incidence of 1.6 per 100,000 and is more common in people in the third to fifth decades of life. The prevalence of cervical disc herniation increases with age in both men and women. It is more common in women and accounts for more than 60% of cases. Cervical disc herniation is a spine disease that seriously affects the quality of life of patients and imposes a heavy economic burden on individuals and society. In recent years, with the widespread use of mobile phones and computers and the increase in the life pressure of today's people, the incidence of cervical disc herniation has shown a younger trend. The role of surgical and non-surgical treatment of patients with cervical disc herniation has not been adequately investigated. While the majority of published data reflects surgical outcomes, there is little data on the outcomes of patients treated without surgery. The most commonly used non-surgical treatments are manipulation, mobilization, kinesiology taping and therapeutic exercises along with electrotherapy agents such as laser therapy, TENS, vacuum interferential and traction. Exercise is considered one of the evidence-based methods to reduce pain in cervical disc herniation, prevent further injury, increase muscle strength, endurance and flexibility, improve proprioception, and contribute to and maintain normal life activities. Exercises used in neck pain in the literature consist of various exercises such as cervical isometrics, cervical concentric/eccentric exercises using pulley systems or weights, upper extremity exercises using dumbbells or deep neck flexor/extensor rehabilitation. Isometric exercises are effective in treating neck pain, range of motion and disability.

DETAILED DESCRIPTION:
It has been reported in the literature that neck stabilization exercises should be included in the rehabilitation of patients with chronic neck pain, as they increase the strength, endurance and coordination of the spinal stabilizer muscles and therefore help in reducing neck pain and improving cervical functions. Cervical stabilization exercises are a method of exercise designed to improve the innate mechanisms that enable the cervical spine to maintain a stable, injury-free state, as in the lumbar spine. Despite the popularity of stabilization exercises, which are performed with a series of exercises that are relatively simple in terms of time and equipment, but physiologically complex, in the treatment of back and pelvic pain, no randomized controlled trial (RCT) has investigated its effectiveness on neck pain, disability, strength, flexibility and quality of life in cases with cervical disc herniation. There is a deficiency.

Therefore, in this study, investigators aim to evaluate and compare the effectiveness of three-week cervical stabilization exercises and cervical isometric exercises on neck pain, disability, strength, flexibility and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Cervical Disc Herniation
2. Complaints started at least 3 months ago
3. Patients with cervical disc herniation between the ages of 18-60;
4. Has not received physical therapy or rehabilitation in the last 3 months;
5. Not taking any medication such as analgesics, anti-inflammatory drugs or muscle relaxants to treat the symptoms.

Exclusion Criteria:

1. major psychiatric illness,
2. Patients with cervical spine surgery and rheumatological diseases;
3. pacemaker users;
4. Those who are injected with local corticosteroids;
5. pregnant woman; Cancer patients.
6. Patients who refuse to participate in the study will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Visual analog Scale (VAS) | 3 weeks
  A visual analog scale (VAS) will be used to evaluate the patient's pain intensity. Patients will be asked to describe their current pain by marking "no pain" and "worst possible pain" on a 100 mm horizontal line.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | 3 weeks
  The Neck Disability Index (NDI) is a 10-item questionnaire that measures self-reported disability related to neck pain. The NDI is the most widely used, translated, and oldest questionnaire for neck pain. It has been shown to have high "test-retest" reliability. The NDI has also been shown to be valid when compared to other measures of pain and disability.
Universal Goniometer | 3 weeks
  Cervical Joint range of motion will be measured using a Universal goniometer (UG). Universal goniometer is a reliable device to evaluate Cervical ROM (3). For measurement of cervical ROM, after the subjects are seated sideways on the physiotherapist, the pivot point will be placed on the lateral projection of the acromion, measurements will be made while the fixed arm of the goniometer is kept parallel to the ground and the movable arm of the goniometer follows the midline during movement.
Manual Muscle testing | 3 weeks
  Manual muscle testing (MMT) is scored using the 0-5 point Medical Research Council muscle strength rating scale and is a common method of assessing muscle strength in therapeutic trials. MMT is less time consuming and MMT's rating system is subjective.
SF 12 (Short Form 12) | 3 weeks
  SF-12, a measure of Health-Related Quality of Life, can be used in age, disease and treatment groups. It is a shortened version of the SF-36 and contains 12 questions, each with two to five answer options. The patient is told to choose the option that best suits him/her. The SF-12 covers eight dimensions: general health, physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. A physical and mental health score, each ranging from 0 to 100, can be calculated using scoring algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Ozaras, Professor, Study Chair — Uskudar University, Faculty of Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - NPIstanbul Brain Hospital, Istanbul
  - Uskudar University NPIstanbul Brain Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No
After I complete my study I will decide to share.

REFERENCES:
- [Background] Yoon WW, Koch J. Herniated discs: when is surgery necessary? EFORT Open Rev. 2021 Jun 28;6(6):526-530. doi: 10.1302/2058-5241.6.210020. eCollection 2021 Jun. PMID 34267943
- [Background] Wong JJ, Cote P, Quesnele JJ, Stern PJ, Mior SA. The course and prognostic factors of symptomatic cervical disc herniation with radiculopathy: a systematic review of the literature. Spine J. 2014 Aug 1;14(8):1781-9. doi: 10.1016/j.spinee.2014.02.032. Epub 2014 Mar 12. PMID 24614255
- [Background] Xu Q, Tian X, Bao X, Liu D, Zeng F, Sun Q. Nonsurgical spinal decompression system traction combined with electroacupuncture in the treatment of multi-segmental cervical disc herniation: A case report. Medicine (Baltimore). 2022 Jan 21;101(3):e28540. doi: 10.1097/MD.0000000000028540. PMID 35060512
- [Background] Saal JS, Saal JA, Yurth EF. Nonoperative management of herniated cervical intervertebral disc with radiculopathy. Spine (Phila Pa 1976). 1996 Aug 15;21(16):1877-83. doi: 10.1097/00007632-199608150-00008. PMID 8875719
- [Background] Yilmaz M, Tarakci D, Tarakci E. Comparison of high-intensity laser therapy and combination of ultrasound treatment and transcutaneous nerve stimulation on cervical pain associated with cervical disc herniation: A randomized trial. Complement Ther Med. 2020 Mar;49:102295. doi: 10.1016/j.ctim.2019.102295. Epub 2020 Jan 3. PMID 32147037
- [Background] Celenay ST, Kaya DO, Akbayrak T. Cervical and scapulothoracic stabilization exercises with and without connective tissue massage for chronic mechanical neck pain: A prospective, randomised controlled trial. Man Ther. 2016 Feb;21:144-50. doi: 10.1016/j.math.2015.07.003. Epub 2015 Jul 15. PMID 26211422
- [Background] Price J, Rushton A, Tyros I, Tyros V, Heneghan NR. Effectiveness and optimal dosage of exercise training for chronic non-specific neck pain: A systematic review with a narrative synthesis. PLoS One. 2020 Jun 10;15(6):e0234511. doi: 10.1371/journal.pone.0234511. eCollection 2020. PMID 32520970
- [Background] Dusunceli Y, Ozturk C, Atamaz F, Hepguler S, Durmaz B. Efficacy of neck stabilization exercises for neck pain: a randomized controlled study. J Rehabil Med. 2009 Jul;41(8):626-31. doi: 10.2340/16501977-0392. PMID 19565156
- [Background] Kuo YL, Lee TH, Tsai YJ. Evaluation of a Cervical Stabilization Exercise Program for Pain, Disability, and Physical Impairments in University Violinists with Nonspecific Neck Pain. Int J Environ Res Public Health. 2020 Jul 28;17(15):5430. doi: 10.3390/ijerph17155430. PMID 32731521
- [Background] Avaghade RR, Shinde SB, Dhane SB. Effectiveness of McKenzie approach and segmental spinal stabilization exercises on neck pain in individuals with cervical postural syndrome: An experimental study. J Educ Health Promot. 2023 Jul 29;12:225. doi: 10.4103/jehp.jehp_239_23. eCollection 2023. PMID 37727425
- [Background] Sadeghi A, Rostami M, Ameri S, Karimi Moghaddam A, Karimi Moghaddam Z, Zeraatchi A. Effectiveness of isometric exercises on disability and pain of cervical spondylosis: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2022 Jun 16;14(1):108. doi: 10.1186/s13102-022-00500-7. PMID 35710510